CLINICAL TRIAL: NCT07122479
Title: Prevention of Hospital Acquired Deconditioning in Hospitalized Acute Leukemia Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-0527
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-Prong Approach to Reduce Hospital Acquired Deconditioning (Other): The intervention is a three-prong approach to reduce hospital acquired deconditioning in patients with anticipated prolonged length of stay for acute leukemia chemotherapy. The intervention includes 1) providing and demonstrating a set of daily physical exercises to patient according to their baseline performance status as assessed by physical therapist, 2) maintaining a patient-completed daily log of physical exercise adherence and 3) standardize the monitoring of physical exercise by the healthcare team by its inclusion in daily progress notes.
  Interventions: Other: Three-Pronged Approach to Reduce Hospital Acquired Deconditioning

INTERVENTIONS:
Other: Three-Pronged Approach to Reduce Hospital Acquired Deconditioning — The intervention includes 1) providing and demonstrating a set of daily physical exercises to patient according to their baseline performance status as assessed by physical therapist, 2) maintaining a patient-completed daily log of physical exercise adherence and 3) standardize the monitoring of physical exercise by the healthcare team by its inclusion in daily progress notes.

SUMMARY:
This study aims to decrease the incidence of hospital acquired deconditioning (HAD) and to help standardize daily physical exercise monitoring in acute leukemia patients with anticipated prolonged duration of hospital stay. The investigators hypothesize that implementing a patient-reported adherence log of their recommended standard daily set of exercises will help reduce proportion of hospital acquired deconditioning in acute leukemia patients. The investigators also hypothesize that less adherent patients will have more inpatient hospital related events and decreased health related quality of life.

DETAILED DESCRIPTION:
Hospital-associated deconditioning (HAD), or post-hospital syndrome, describes the physical, cognitive, and functional decline that develops during hospitalization. Acute leukemia patients require inpatient chemotherapy treatments that often impose a minimal hospital stay of 21 days. While physical activity is recommended, its prescription and monitoring are not standardized, often leading to deconditioning developing before physical activity is urged.

This study aims to decrease the incidence of hospital acquired deconditioning (HAD) and to help standardize daily physical exercise monitoring in acute leukemia patients with anticipated prolonged duration of hospital stay. The investigators hypothesize that implementing a patient-reported adherence log of their recommended standard daily set of exercises will help reduce proportion of hospital acquired deconditioning in acute leukemia patients. The investigators also hypothesize that less adherent patients will have more inpatient hospital related events and decreased health related quality of life.

The intervention is a three-prong approach to reduce hospital acquired deconditioning in patients with anticipated prolonged length of stay for acute leukemia chemotherapy at North Shore University Hospital. The intervention includes 1) providing a set of daily physical exercises to patient according to their baseline performance status as assessed by physical therapist, 2) maintaining a patient-completed daily log of physical exercise adherence and 3) standardize the monitoring of physical exercise by the healthcare team by its inclusion in daily progress notes.

The results will assess the effectiveness of this intervention in reducing the occurrence proportion of HAD in the intervention group compared to historical controls. Additionally, the investigators will assess the correlation between patient reported adherence rate to the occurrence of hospital related events as well as its impact on health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99
* Patient admitted to North Shore University Hospital on 7Monti floor
* Diagnosis of acute leukemia (AML or ALL)
* Admitted for treatment with remission inducing therapy either in frontline, relapsed or salvage setting with anticipated hospital length of stay of at least 10 days
* ECOG 0-3 on day of induction.

Exclusion Criteria:

* Patients admitted for >14 days prior to initiation of treatment.
* Baseline altered mental status defined by Glasgow coma scale with score less than 15, that does not resolve within first 7 days of treatment as this would preclude participation in physical activity program.
* Baseline disability that would prevent participation in physical activity program.
* CML in acute blast phase.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Assess Effectiveness of Prescribed Physical Exercise Program | 12 months
  daily log of physical exercise adherence and 3) standardize the monitoring of physical exercise by the healthcare team by its inclusion in daily progress notes.

SECONDARY OUTCOMES:
assess the correlation between patient-reported adherence rate (%) of daily physical exercise | 12 months
  to assess the correlation between patient-reported adherence rate (%) of daily physical exercise to occurrence of hospital related events and impact on health-related quality of life.

OTHER OUTCOMES:
Adherence rates of daily physical exercise | 12 months
  To assess if there is a difference in adherence rates of daily physical exercise between age groups
Number of days admitted prior to initiation of treatment | 12 months
  To assess if number of days admitted prior to initiation of treatment affects adherence rates to daily physical activity
Impact of adherence to daily physical activity on re-admission rates | 12 months
  To assess the impact of adherence to daily physical activity on re-admission rates for complications within 6 months of induction treatment
Assess impact of adherence to daily physical activity on hospital admission cost | 12 months
  To assess impact of adherence to daily physical activity on hospital admission cost
Assess if daily recording of physical activity improves monitoring | 12 months
  To assess if daily recording of physical activity improves monitoring of risk for HAD

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Boisclair, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital (NSUH), Manhasset, New York
  - Zuckerberg Cancer Center, New Hyde Park, New York

IPD SHARING:
Plan to Share IPD: No